CLINICAL TRIAL: NCT01249807
Title: Taiwanese People's Willingness to Participate in Cancer Screening: Colon, Oral Cavity, Breast, and Cervical Cancer Screening
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: China Medical University Hospital, China Medical University Hospital
Other Study IDs: DMR99-IRB-185
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
Keywords: Cancer Screening; health service utilization model; quality of health life

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Patients, Family, Community member

SUMMARY:
Cancer Screening is necessary for promoting cancer prevention in the area of public health. The Department of Health, Executive Yuan of the Republic of China has expanded and included colon cancer screening, oral cavity cancer screening, breast cancer screening, and cervical cancer screening in national-wide preventive healthcare services. However, most of the Taiwanese do not have the concepts of what cancer screening is and regular participation of cancer screening. This will easily cause their neglect of quality of personal healthcare and habits of cancer screening. Recently, in order to reach the national goal of cancer prevention, the parallel methods, multi-promotion for reinforcing concepts and free cancer screening, have been utilized to cultivate Taiwanese people's active participation of cancer screening. Therefore, this study will use health service utilization model to investigate Taiwanese people's concepts of cancer-related knowledge and the major causes of low participation of cancer screening.

In order to investigate Taiwanese people's health service utilization model and quality of health life, this study first review the related regulations and screening rates of cancer prevention, including cancers of colon, oral cavity, breast, and cervical, in Taiwan. In addition, the structured questionnaire will be conducted to collect, investigate, and analyze the relationship between the willingness of participating the aforementioned cancer screening and personal characteristics, quality of health life, medical history, and concepts of cancer, etc. It is expected that the results of this study will provide accurate and effective promotions of cancer screening to medical institutions and medical affairs to reinforce the concepts of participation for raising the rates of cancer screening; furthermore, to awaken Taiwanese people's crucial awareness of early treatment improves the chances of recovery on cancer.

ELIGIBILITY:
Inclusion Criteria:

Cases who are willing to answer the questionnaire

Exclusion Criteria:

Cases who are not willing to answer the questionnaire

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients patients' families Community people
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-10 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taichung, Taiwan